CLINICAL TRIAL: NCT01316666
Title: Norepinephrine Transporter Blockade as a Pathophysiological Biomarker in Neurogenic Orthostatic Hypotension
Brief Title: Norepinephrine Transporter Blockade as a Pathological Biomarker in Neurogenic Orthostatic Hypotension
Acronym: 6103
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Italo Biaggioni, MD, Vanderbilt University
Other Study IDs: 101311; U54NS065736 (NIH)
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Orthostatic Hypotension; Pure Autonomic Failure; Multiple System Atrophy; Parkinson's Disease
Keywords: orthostatic hypotension; Multiple System Atrophy; Pure Autonomic Failure; Parkinson's Disease
MeSH Terms: conditions — Hypotension, Orthostatic; Pure Autonomic Failure; Multiple System Atrophy; Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neurogenic Hypotension: Patients with neurogenic hypotension, which includes those with Pure Autonomic Failure (PAF), Multiple System Atrophy (MSA) and Parkinson Disease (PD)

SUMMARY:
The autonomic or automatic nervous system helps control blood pressure. Diseases of the autonomic nervous system may result in a drop in blood pressure on standing in many cases leading to fainting. Diseases that affect the autonomic nervous system include pure autonomic failure, multiple system atrophy and Parkinson's disease, and can present with very similar symptoms and it is sometimes difficult to determine an exact diagnosis. The purpose of the study is to find out if the blood pressure response from taking a single dose of the medication atomoxetine can help in the diagnosis of these diseases.

DETAILED DESCRIPTION:
This is an observational, prospective three-year longitudinal study. The investigators will enroll participants with primary neurogenic orthostatic hypotension. All participants will undergo an extensive neurological and cardiovascular evaluation, including detailed autonomic testing and quality of life assessment. The investigators will then determine the magnitude of the pressor effect produced by 18 mg atomoxetine given orally, measured 1 hour after drug administration. Participants will be followed annually or more often if there is a significant change in their clinical condition. During follow up at year 3, the investigators will repeat the initial neurological, cardiovascular and autonomic evaluation. The primary endpoint would be the final diagnosis made at year 3 after the initial evaluation (at the end of the follow-up period) or if they develop significant worsening of symptoms during follow-up phone assessments, based on specific clinical criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old with Neurogenic orthostatic hypotension, ≥30 mmHg drop in SBP within 5 minutes of standing
* Associated with impaired autonomic reflexes, as determined by absence of blood pressure overshoot during phase IV of the Valsalva maneuver
* Absence of other identifiable causes of autonomic neuropathy
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnancy
* Systemic illnesses known to produce autonomic neuropathy, including but not limited to diabetes mellitus, amyloidosis, monoclonal gammopathy of unknown significance, and autoimmune neuropathies
* Known intolerance to atomoxetine, Pre-existing sustained severe hypertension (BP at least 180/110 mmHg in the sitting position)
* Clinically unstable coronary artery disease, or major cardiovascular or neurological event in the past 6 months
* Any other significant systemic, hepatic, cardiac or renal illness
* Use of MAO-I within 14 days
* Known closed-angle glaucoma or Life-threatening arrhythmias

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants with neurogenic orthostatic hypotension, which is a drop in systolic blood pressure of at least 30 mmHg within 5 minutes of standing with associated impaired autonomic reflexes.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Final Diagnosis (pre vs post ganglionic autonomic failure) based on clinical criteria. | 3 years
  Probable MSA - PAF with urinary incontinence or an orthostatic decrease of 30 mmHG in systolic blood pressure within 3 minutes of standing and poorly levodopa responsive parkinsonism or a cerebellar syndome.
  For Possible MSA - parkinsonism or a cerebellar syndrome and one additional feature.
  Probable PAF - orthostatic hypotension and impaired autonomic reflexes in the absence of clinical signs or symptoms of neurodegeneration.
  For Parkinson's Disease: diagnosed based on the United Kingdom Parkinson Disease Society Brain Bank clinical diagnostic criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center (Harvard), Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - New York University, New York, New York
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Background] Birkenfeld AL, Schroeder C, Boschmann M, Tank J, Franke G, Luft FC, Biaggioni I, Sharma AM, Jordan J. Paradoxical effect of sibutramine on autonomic cardiovascular regulation. Circulation. 2002 Nov 5;106(19):2459-65. doi: 10.1161/01.cir.0000036370.31856.73. PMID 12417543
- [Background] Esler MD, Wallin G, Dorward PK, Eisenhofer G, Westerman R, Meredith I, Lambert G, Cox HS, Jennings G. Effects of desipramine on sympathetic nerve firing and norepinephrine spillover to plasma in humans. Am J Physiol. 1991 Apr;260(4 Pt 2):R817-23. doi: 10.1152/ajpregu.1991.260.4.R817. PMID 2012253
- [Background] Gilman S, Low P, Quinn N, Albanese A, Ben-Shlomo Y, Fowler C, Kaufmann H, Klockgether T, Lang A, Lantos P, Litvan I, Mathias C, Oliver E, Robertson D, Schatz I, Wenning G. Consensus statement on the diagnosis of multiple system atrophy. American Autonomic Society and American Academy of Neurology. Clin Auton Res. 1998 Dec;8(6):359-62. doi: 10.1007/BF02309628. PMID 9869555
- [Background] Gilman S, Wenning GK, Low PA, Brooks DJ, Mathias CJ, Trojanowski JQ, Wood NW, Colosimo C, Durr A, Fowler CJ, Kaufmann H, Klockgether T, Lees A, Poewe W, Quinn N, Revesz T, Robertson D, Sandroni P, Seppi K, Vidailhet M. Second consensus statement on the diagnosis of multiple system atrophy. Neurology. 2008 Aug 26;71(9):670-6. doi: 10.1212/01.wnl.0000324625.00404.15. PMID 18725592
- [Background] Goldstein DS, Holmes C. Metabolic fate of the sympathoneural imaging agent 6-[18F]fluorodopamine in humans. Clin Exp Hypertens. 1997 Jan-Feb;19(1-2):155-61. doi: 10.3109/10641969709080812. PMID 9028643
- [Background] Goldstein DS, Polinsky RJ, Garty M, Robertson D, Brown RT, Biaggioni I, Stull R, Kopin IJ. Patterns of plasma levels of catechols in neurogenic orthostatic hypotension. Ann Neurol. 1989 Oct;26(4):558-63. doi: 10.1002/ana.410260410. PMID 2510587
- [Background] Horimoto Y, Matsumoto M, Akatsu H, Ikari H, Kojima K, Yamamoto T, Otsuka Y, Ojika K, Ueda R, Kosaka K. Autonomic dysfunctions in dementia with Lewy bodies. J Neurol. 2003 May;250(5):530-3. doi: 10.1007/s00415-003-1029-9. PMID 12736730
- [Background] Kaufmann H, Nahm K, Purohit D, Wolfe D. Autonomic failure as the initial presentation of Parkinson disease and dementia with Lewy bodies. Neurology. 2004 Sep 28;63(6):1093-5. doi: 10.1212/01.wnl.0000138500.73671.dc. PMID 15452307
- See also: Beth Israel Deaconess Medical Center Department of Neurology — http://www.bidmc.org/CentersandDepartments/Departments/Neurology.aspx